CLINICAL TRIAL: NCT03288792
Title: A Prospective Multicenter Evaluation of Three Dimensional Functional Metabolic and Risk Assessment System in Women With Mammographically Dense Breasts
Brief Title: A Evaluation of 3D Functional MIRA System in Women With Mammographically Dense Breasts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision, not safety related
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 960-CSP-USA_DenseBreasts_USS1
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RI8 device imaging (Experimental): RI8 Device imaging for adjunctive detection of breast cancer
  Interventions: Device: RI8 device imaging

INTERVENTIONS:
Device: RI8 device imaging — RI8 Device imaging for adjunctive detection of breast cancer
  Other Names: Real Imager 8

SUMMARY:
The purpose of this image acquisition study is to compare, in a Reader Study, the RI8 system used in conjunction with a conventional mammography to mammography alone, and to determine whether the addition of supplementary RI8 result will improve ROC area under the curve. The study is prospective, multi-center, sequential, control trial with the woman serving as her own control. Women determined to have heterogeneously or extremely dense breast based on her previous mammogram and are undergoing routine screening mammography at one of the clinical sites assigned for this study will be eligible to join the study.

ELIGIBILITY:
Inclusion Criteria:

A. Subjects whose most recent (within 18 months) prior mammogram interpreted as heterogeneously dense (ACR BI-RADS Breast Density C) or extremely dense (ACR BI-RADS Breast Density D) breast tissue.

AND

B. Subjects who are asymptomatic and scheduled to undergo routine screening mammography.

OR

C. Subjects scheduled for image-guided needle biopsy as a result of findings obtained during standard of care imaging modalities (mammography, ultrasound and/or MRI) performed at the clinical site that participates in the study.

Exclusion Criteria:

1. Male by birth.
2. Individual is less than 40 and greater than 70 years old.
3. Contraindication to bilateral mammography or MRI.
4. Subjects who are unable to read, understand and execute the informed consent procedure.
5. Subjects who have had mammography, ultrasound or MRI examination performed on the day of the study prior to RI8 scan.
6. Subjects who are pre-menopausal and are between the 14th and 28th day after the start of the menstrual cycle
7. Subjects who have significant existing breast trauma.
8. Subjects who have undergone lumpectomy/mastectomy.
9. Subjects who have undergone breast reduction or breast augmentation.
10. Subjects who have undergone any other type of breast surgery, including surgical biopsy.
11. Subjects who have large breast scar / breast deformation
12. Subjects who have undergone a breast needle biopsy within the 6-week period prior to their intended enrollment into the study.
13. Subjects who have a temperature > 100° F (37.8C) degrees on the day of the RI8 imaging.
14. Subjects who are pregnant or lactating.
15. Subjects with known Raynaud's Disease.
16. Subjects with known Mastitis.
17. Subjects diagnosed with epileptic seizures.
18. Subjects with weight > 135kg (~300 Lbs.).
19. Subjects who are claustrophobic or have physical limitations that do not allow them to sit in the system chair for the required imaging session.
20. Subjects with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices.
21. Subject with kidney failure
22. Subject with known allergy to gadolinium
23. Subject with a history of multiple contrast MRI scans (more than 4 MRI scans over the past two year)
24. Inmates (45 CFR 46.306) or mentally disabled individuals.
25. Subjects with a BI-RADS category 6 (e.g. for which mammogram was performed for the purpose of planning cancer therapy).
26. Subjects currently participating in another investigational clinical study.
27. Subject scheduled for a biopsy due to suspicious symptomatic lump
28. Subjects who participated in the Validation Phase will not be able to participate in the Testing Phase

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in the area under the ROC curve when comparing mammography plus RI8 result to mammography alone. | 18 months
All adverse events and serious adverse events caused by the imaging session as judged by the physician. | 18 months

SECONDARY OUTCOMES:
Sensitivity and specificity will be computed based on the forced BI-RADS assessment of each mammography case alone and mammography plus RI8. | 18 months

OTHER OUTCOMES:
Sensitivity and specificity of the device will be determined from all enrolled cases. Upper and lower estimates will be determined based on missing data. | 18 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Saddleback MemorialCare Breast Center, Laguna Hills, California
  - Memorial Healthcare System, Hollywood, Florida
  - Doris Shaheen Breast Health Center Piedmont Hospital, Atlanta, Georgia
  - The Jackson Clinic, Jackson, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Web site — http://www.realimaging.com